CLINICAL TRIAL: NCT06923202
Title: Study of Alloknesia in Atopic Dermatitis
Acronym: ALLOKNESIE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Collaborators: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0355
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatosis; Alloknesie

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with atopic dermatitis: Patients will take part in the study on a single occasion, during which they will complete the various questionnaires (Alloknesia diagnostic questionnaire, WI-NRS scale, ItchyQol questionnaire, DLQI questionnaire, HADS questionnaire, PUSH-D questionnaire, PSS (Perceived Stress Scale), Epworth questionnaire, ISS questionnaire). There will be no follow-up.

SUMMARY:
Alloknesia is defined as pruritus (= itching) triggered by light mechanical stimuli, which are responsible for the perception of light touch under physiological conditions, but which are perceived as pruritic under pathological conditions. Alloknesia occurs mainly in the context of chronic pruritus. Consequently, patients suffering from chronic pruritus frequently perceive light touch sensations as pruritic, which can be particularly unpleasant and alter human interactions and quality of life on a daily basis. However, the epidemiology and burden of alloknesia have never been studied, whatever the cause of chronic pruritus.Atopic dermatitis is one of the main diseases causing chronic itching, and patients frequently complain of alloknesia. In this study, the investigators are studying the frequency of alloknesia in patients with atopic dermatitis and measuring the consequences of alloknesia in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* No opposition from the patient
* Diagnosis of atopic dermatitis more than 6 months old

Exclusion Criteria:

* Patients who are physically or mentally unable to complete the questionnaires.
* Patients on systemic treatment for 1 month or more
* Refusal to participate
* Patients under legal protection (guardianship, curatorship)
* Patients under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atopic dermatitis
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-11-26 (Estimated); Study Completion 2026-11-26 (Estimated)

PRIMARY OUTCOMES:
Alloknesia diagnostic questionnaire | At enrollment. If the patient completes the questionnaires at home, they will be brought back by the patient at their next medical consultation.
  The questionnaire consists of a single question: 'Can the touch of your skin by clothing, air movements or the light touch of an object or another person trigger itching?

SECONDARY OUTCOMES:
WI-NRS scale / Worst Itch Numeric Rating Scale | At enrollment. If the patient completes the questionnaires at home, they will be brought back by the patient at their next medical consultation.
  Digital pruritus scale, measuring the worst daily itching intensity 0 to 10. 0: no itching 10: worst itch imaginable
ItchyQoL questionnaire / quality-of life instrument for pruritus | At enrollment. If the patient completes the questionnaires at home, they will be brought back by the patient at their next medical consultation.
  Quality-of life instrument for pruritus Itch-related quality of life 0 to 110
DLQI questionnaire / Dermatology Life Quality Index | At enrollment. If the patient completes the questionnaires at home, they will be brought back by the patient at their next medical consultation.
  Skin-related quality of life 0 to 30
HADS questionnaire / Hospital Anxiety and Depression Scale | At enrollment. If the patient completes the questionnaires at home, they will be brought back by the patient at their next medical consultation.
  The HAD scale is an instrument for screening for anxiety and depressive disorders.
  0 to 21
PUSH-D questionnaire / Patient Unique Stigmatization Holistic tool in dermatology | At enrollment. If the patient completes the questionnaires at home, they will be brought back by the patient at their next medical consultation.
  PUSH-D allows a comprehensive view of the degree of stigmatization in visible skin disorders.
  0 to 68
Stress perçu : PSS / Perceived Stress Scale | At enrollment. If the patient completes the questionnaires at home, they will be brought back by the patient at their next medical consultation.
  The PSS (Perceived Stress Scale) is a scale for measuring perceived stress. 0 to 40
Epworth questionnaire / sleepiness scale | At enrollment. If the patient completes the questionnaires at home, they will be brought back by the patient at their next medical consultation.
  The Epworth Test is a self-administered questionnaire that assesses subjective sleepiness and fatigue.
  0 to 21
ISS questionnaire / Sexual Satisfaction Index | At enrollment. If the patient completes the questionnaires at home, they will be brought back by the patient at their next medical consultation.
  Satisfaction with sexual relations 25 to 175

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU d'Angers, Angers
  - CHU de Brest, Brest
  - CHD Vendée, La Roche-sur-Yon
  - Groupe Hospitalier Bretagne Sud, Lorient
  - CHU de Nantes Hôtel-Dieu, Nantes
  - CHU de Rennes, Rennes
  - CHU de Tours, Tours
  - CH Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Kimel M, Zeidler C, Kwon P, Revicki D, Stander S. Validation of Psychometric Properties of the Itch Numeric Rating Scale for Pruritus Associated With Prurigo Nodularis: A Secondary Analysis of a Randomized Clinical Trial. JAMA Dermatol. 2020 Dec 1;156(12):1354-1358. doi: 10.1001/jamadermatol.2020.3071. PMID 32936233